CLINICAL TRIAL: NCT03177109
Title: Comparison of Fluoride Varnish With Two Different Desensitizers in Reducing Dentinal Hypersensitivity
Brief Title: Comparison of Different Desensitizers in Reducing Dentinal Hypersensitivity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Hasan Hameed, Resident investigator, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 4714-Sur-ERC-17
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Dentine Hypersensitivity
Keywords: Dentine Hypersensitivity; Fluoride varnish; Desensitizing agents
MeSH Terms: conditions — Dentin Sensitivity | interventions — CMW cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Fluoride Varnish Group (Active Comparator): 5% fluoride varnish (Acclean) applied topically
  Interventions: Drug: 5% fluoride varnish
- Arginine paste Group (Active Comparator): 8% arginine containing paste (Colgate® Sensitive Pro-Relief™) applied topically
  Interventions: Drug: 8% arginine containing paste
- Adhesive Resin Group (Active Comparator): Self-adhesive resin (Seal and Protect, Dentsply) applied topically
  Interventions: Drug: Self-adhesive resin

INTERVENTIONS:
Drug: 5% fluoride varnish — Applied topically as a coating at single point in time
  Other Names: Acclean
  Arms: Fluoride Varnish Group
Drug: 8% arginine containing paste — Applied topically as a coating at single point in time
  Other Names: Colgate® Sensitive Pro-Relief™
  Arms: Arginine paste Group
Drug: Self-adhesive resin — Applied topically as a coating at single point in time and light cured for 20 seconds
  Other Names: Seal and Protect, Dentsply
  Arms: Adhesive Resin Group

SUMMARY:
This is a single center, randomized control. Sixty eligible subjects will be recruited into 3 study treatment groups (n=20 per group) through computerized randomization. Subjects in group 1 will be treated with 8% arginine containing paste(Colgate® Sensitive Pro-Relief™), group 2 with 5% topical fluoride varnish (Acclean) and group 3 with self-adhesive resin (Seal and protect, Dentsply). The subjects in the study will be evaluated for tactile and air-blast hypersensitivity criteria at baseline, two and four weeks.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the efficacy of three common professionally applied desensitizing agents in the reduction of dentine hypersensitivity over a period of 4 weeks. Patients presenting to the dental clinic with Dentine hypersensitivity and fulfilling the inclusion criteria will be included in the study after taking informed consent. Participants will be divided into three groups. Sixty eligible subjects will be recruited into 3 study treatment groups (n=20 per group) through computerized randomization. Subjects in group 1 will be treated with 8% arginine containing paste(Colgate® Sensitive Pro-Relief™), group 2 with 5% topical fluoride varnish (Acclean) and group 3 with self-adhesive resin (Seal and protect, Dentsply). the subjects in the study will be evaluated for tactile and air-blast hypersensitivity criteria at baseline, two and at four weeks by another dentist who would be a blind assessor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18 and above with dentine hypersensitivity will be selected.
* At least two hypersensitive teeth which will be sensitive to air blast (Schiff air sensitivity scores of 2 or 3) and positive tactile sensitivity assessed clinically with explorer
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* • Patients who would have undergone any periodontal procedure or gotten any professionally applied desensitizers in the last three months.

  * Patients having generalized sensitivity in all teeth
  * Chronic use of anti-inflammatory and analgesic medications
  * Pregnant or lactating females;
  * Any denture bridgework; active cervical caries or deep abrasion requiring Class V fillings;
  * Fractured, crowned or root filled teeth and teeth with large restorations
  * Carious teeth or cracked teeth assessed on the basis of clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of hypersensitivity | Reduction of hypersensitivity will be assessed at 2 weeks and 4 weeks
  • Investigators are comparing the effectiveness of three professionally applied desensitizing agents, 8% arginine containing paste (Colgate® Sensitive Pro-Relief™), 5% fluoride varnish (Acclean) and self-adhesive resin (Seal and Protect, Dentsply) in reducing the dentine hypersensitivity immediately after application and at 2 and 4 weeks follow-up.The measurements of sensitivity will be determined by patient's response to air blast stimuli. Subjective responses will be recorded using Schiff Cold Air Sensitivity Scale which is scored as follows:
  0 Subject does not respond to air stimulus,
  1. Subject responds to air stimulus but does not request discontinuation of stimulus
  2. Subject responds to air stimulus and requests discontinuation or moves from stimulus
  3. Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan Hameed, BDS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No